CLINICAL TRIAL: NCT01785992
Title: A Phase II Study to Assess the Safety and Efficacy of the Steroid Sulfa-tase Inhibitor Irosustat When Added to an Aromatase Inhibitor in ER Positive Locally Advanced or Metastatic Breast Cancer Patients.
Brief Title: A Study of the Safety and Effectiveness of Irosustat When Added to an AI in ER+ve Locally Advanced or Metastatic Breast Cancer.
Acronym: IRIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C/22/2011; 2011-005680-25 (EudraCT Number)
Record Dates: First submitted 2013-02-04; First posted 2013-02-07 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2014-03

CONDITIONS: Locally Advanced Breast Cancer; Metastatic Breast Cancer
Keywords: Oestrogen receptor; Locally advanced; Metastatic; Breast cancer; Sulfatase inhibitor
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — irosustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Irosustat (Single arm study) (Other): Patients will receive 40mg of Irosustat once daily in addition to the aromatase inhibitor on which they progressed until disease progression or the development of unacceptable toxicities.
  Interventions: Drug: Irosustat

INTERVENTIONS:
Drug: Irosustat — Patients will receive 40mg of Irosustat once daily in addition to the aromatase inhibitor on which they progressed until disease progression or development of unacceptable toxicities.
  Other Names: STX64; 667 Coumate; BN83495

SUMMARY:
70% of breast cancers that occur in postmenopausal women rely on the hormone oestrogen to grow and are likely to respond to hormone treatment. This type of treatment reduces the amount of oestrogen in the body, slowing the growth of cancer or stopping it altogether. One type of hormone treatment, aromatase inhibitors (AIs), works by stopping the body from making oestrogen. Currently, women with locally advanced or metastatic breast cancer that is not being controlled by one class of AI are switched to the other class of AI. The reason for this is that some cancer cells can become resistant to one class but are still sensitive to the other class. However, oestrogen can be made in the body by two pathways and AIs block only one of these pathways. A new drug called Irosustat can reduce the production of oestrogen in the body by blocking the second pathway. This study is investigating whether adding Irosustat to AI treatment i.e. blocking both pathways at the same time, can further reduce the amount of oestrogen in the body and therefore control the breast cancer better.

27 postmenopausal women with oestrogen receptor positive locally advanced or metastatic breast cancer that is not being controlled by their current AI treatment will be recruited in this study from 9 United Kingdom (UK) hospitals. Eligible patients will receive 40mg of Irosustat once daily in addition to the AI on which they progressed. Patients will receive Irosustat for as long as it controls their cancer or until they have side effects that stop them from taking treatment. Patients will be seen monthly for the first 6 months and every 3 months thereafter. Participating patients will also be given the option to take part in the exploratory part of this study by donating tissue and blood samples.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to admission to this study.
2. Aged ≥ 25 years of age.
3. Histologically confirmed ER+ve primary or metastatic breast cancer.
4. Locally advanced or metastatic breast cancer treated with 1st line AI treatment with either a documented objective response (CR/PR) or disease stabilisation (SD) for at least 6 months prior to disease progression.
5. Postmenopausal as defined by any of the following criteria:

   1. Amenorrhoea for at least 6 months prior to study entry and estradiol and LH/FSH in the postmenopausal range on local laboratory analysis whilst taking a 3rd generation AI during the screening phase of the study.
   2. Amenorrhoea during combination treatment with ovarian suppression (e.g. goserelin) and an AI in which case estradiol should be below the limit of detection of the standard local laboratory assay during the screening phase of the study.
6. ECOG performance status 0 to 2.
7. Measurable and/or evaluable sites of locally advanced or metastatic disease that can be accurately assessed by CT/MRI scan at baseline and follow up visits (RECIST v1.1).

   N.B Patients with bone metastasis are eligible provided they have evaluable metastases sites that can be followed (X-Ray or MRI/CT scanning). Patients on established bisphosphonate treatment for at least 3 months are eligible for entry into the trial and are allowed to continue with bisphosphonate treatment.
8. Adequate organ function as defined by (Haemoglobin (Hb) ≥ 9 g/dL; Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L; Platelet count (Plts) ≥ 100 ≥ 109/L; White Blood Cell (WBC) ≥ 3.0 x 109/L; Serum albumin ≤ 1.5 upper limit of normal (ULN); Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤ 3 x ULN if no demonstrable liver metastases or ≤ 5 x ULN in the presence of liver metastases; alkaline phosphatase (ALP) ≤ 5 x ULN; Total bilirubin ≤ 1.5 x ULN if no demonstrable liver metastases or ≤ 3 x ULN in the presence of liver metastases; Creatinine ≤ 1.5 x ULN or creatinine clearance >50ml/min).
9. Life expectancy of ≥3 months.

Exclusion Criteria:

1. Human epidermal growth factor Receptor-2 (HER2) positive cancer.
2. Discontinuation of current AI therapy for > 21 days prior to study entry.

   N.B If the patient has discontinued the AI within this period they can be restarted on the same AI. This must be continued for at least 7 days before introducing the IMP. Baseline investigations must be performed in timeframes related to the start of the IMP, not the AI.
3. Rapidly progressive, life-threatening metastases, including any of the following:

   1. Patients with active parenchymal brain or leptomeningeal involvement
   2. Symptomatic lymphangitis carcinomatosis
   3. Extensive visceral metastases requiring chemotherapy.
4. Patients with a history of another primary malignancy within 5 years prior to starting study treatment, except adequately treated basal or squamous cell carcinoma of the skin, carcinoma in site and the disease under study.
5. More than one prior line of chemotherapy for locally advanced or metastatic disease.
6. AI therapy given in combination with another endocrine agent with the exception of a GnRH agonist.
7. Radiotherapy to measurable lesion within 2 months of treatment start.
8. Systemic corticosteroids for ≥ 15 days within the last 4 weeks.
9. Evidence of uncontrolled active infection.
10. Evidence of significant medical condition or laboratory finding which, in the opinion of the Investigator, makes it undesirable for the patient to participate in the trial.
11. Concurrent therapy with any other investigational agent.
12. Concomitant use within 14 days prior to commencement of study treatment of:

    1. Rifampicin and other CYP2C and 3A inducers such as rifabutin, rifapentine, carbamazepine, phenobarbital, phenytoin and St. John's Wort
    2. Systemic carbonic anhydrase inhibitors.
13. Any of the following cardiac criteria:

    1. Mean resting corrected QT interval (QTcf) >450 ms as calculated by Fridericia's formula obtained from 3 electrocardiograms (ECGs)
    2. Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG e.g. complete left bundle branch block, third degree heart block
    3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age or any concomitant medication known to prolong the QT interval.
14. Uncontrolled abnormalities of serum potassium, sodium, calcium (corrected) phosphate or magnesium levels.
15. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated investigational medicinal product (IMP) or previous significant bowel resection that would preclude absorption of Irosustat or the AI.

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Clinical benefit defined as complete response / partial response plus stable disease for at least 6 months (RECIST v1.1). | Patients will be followed up until disease progression, an expected average of 6 months

SECONDARY OUTCOMES:
Duration of clinical benefit as defined by the number of days from start of study drug to the first evidence of disease progression or death due to any cause (RECIST v1.1). | Patients will be followed up until disease progression, an expected average of 6 months
Progression Free Survival defined as time from randomisation to first evidence of disease progression or death due to any cause (RECIST v1.1). | Patients will be followed up until disease progression, an expected average of 6 months
Safety and tolerability as assessed by the collection of adverse events according to the Common Terminology Criteria for Adverse Events (CTCAE v 4.03). | Patients will be followed up until disease progression, an expected average of 6 months
To measure alterations in circulating steroid hormones and correlation of these measures with clinical outcome. | 0,1,2,3,4,5,6,9,12 months after study entry
Objective response rate as defined by complete response and partial response (RECIST v1.1) | Patients will be followed up until disease progression, an expected average of 6 months

OTHER OUTCOMES:
To assess tumour proliferation using Ki67 in tumour biopsies taken from the primary and locally advanced or metastatic tumour. | At the time of surgery for primary disease and surgery or biopsy for metastatic disease
To determine the intratumoural expression of ERα and known ERα regulated genes. | At the time of surgery or biopsy of metastatic disease
To determine the expression of steroidogenic enzymes i.e. STS, aromatase, oestrogen sulfotransferase (EST)and 17bHSD1. | At the time of surgery or biopsy of metastatic disease
To collect and store blood samples, archival tumour samples and locally advanced or meta-static tumour samples and analyse surplus blood or tissue for factors that may affect response to Irosustat when given in addition to an AI. | 0,1,2,3,4,5,6,9,12 months after study entry

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Palmieri, Principal Investigator — Imperial College London
Locations (9):
- United Kingdom (9):
  - Mid Essex Hospital Services NHS Trust, Chelmsford
  - NHS Lothian, Edinburgh
  - NHS Greater Glasgow and Clyde, Glasgow
  - Royal Liverpool and Broadgreen University Hospital, Liverpool
  - Royal Free London, London
  - West Middlesex University Hospital NHS Trust, London
  - Imperial College Healthcare NHS Trust, London
  - University College London Hospitals NHS Foundation Trust, London
  - The Christie NHS Foundations Trust, Manchester